CLINICAL TRIAL: NCT02846831
Title: An Open-label, Randomized, Two-way, Cross-over Study to Assess the Efficacy of Single-hormone Closed-loop Strategy and Sensor-augmented Pump Therapy in Regulating Glucose Levels for 12 Days in Free-living Outpatient Conditions in Patients With Type 1 Diabetes
Brief Title: Closed-loop Control of Glucose Levels (Artificial Pancreas) for 12 Days in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-14
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Artificial pancreas; Closed-loop system; Hypoglycemia; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Methods; Insulin Infusion Systems; Continuous Glucose Monitoring; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensor-augmented pump therapy (Active Comparator): Participants will use sensor-augmented pump therapy with low-glucose suspend to regulate glucose levels. The low-glucose suspend feature available in the MiniMed® Paradigm® Veo™, Medtronic combined with the Enlite sensor® will be used. This feature allows for suspension of insulin delivery at a pre-set sensor glucose value for up to 2 hours.
  Interventions: Other: 12-day intervention with sensor-augmented pump therapy; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Insulin
- Single-hormone closed-loop strategy (Active Comparator): Variable subcutaneous insulin infusion will be used to regulate glucose levels. Participant's usual fast-acting insulin analog will be infused using a subcutaneous infusion pump (MiniMed® Paradigm® Veo™, Medtronic). Every 10 minutes, the glucose levels as measured by the sensor (Enlite sensor®, Medtronic) will be transferred automatically to a smartphone, that harbors the algorithm, that will calculate the recommended doses and will send it wirelessly to the infusion pump.
  Interventions: Other: 12-day intervention with single-hormone closed-loop strategy; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Insulin

INTERVENTIONS:
Other: 12-day intervention with sensor-augmented pump therapy — A sensor will be inserted on the day before the start of the intervention by the participants. The participant will also have to install the study insulin pump. Participants will be advised to continue with study intervention at home for the next 12 days.
  Participants will have been previously shown how to use the study insulin pump.
  Arms: Sensor-augmented pump therapy
Other: 12-day intervention with single-hormone closed-loop strategy — A sensor will be inserted on the day before the start of the intervention by the participants. On the first day of the intervention, participants will be admitted to the clinical research facility anytime between 8:00 am and 11:30 am. Training on connection and disconnection of the system, meal boluses, etc. will be given.
  Only participants demonstrating competency on use of study devices will be allowed to continue to the home study phase. Participants will be advised to continue with study intervention at home for the next 12 days.
  Arms: Single-hormone closed-loop strategy
Device: Insulin pump — Tandem Diabetes Care
Device: Continuous glucose monitoring system — Dexcom G5 Platinum
Drug: Insulin — Participant's usual fast-acting insulin analog will be used: Lispro (Humalog), Aspart (NovoRapid) or Glulisine (Apidra)

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings.

The objective of this study is to compare the effectiveness of single-hormone closed-loop and sensor-augmented pump therapy in regulating day-and-night glucose levels in adults with T1D for 12 days in outpatient settings.

The investigators hypothesize that dual-hormone closed-loop will increase the percentage of time of glucose levels spent in the target range in adults compared to single-hormone closed-loop, which in turn will be more effective than sensor-augmented pump therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. HbA1c ≤ 12%.

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator
2. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery
3. Warfarin chronic treatment if INR monitoring cannot be evaluated (can increase the risk of bleeding)
4. Chronic use of acetaminophen. Acetaminophen may interfere with glucose sensor readings
5. Pregnancy (ongoing or current attempt to become pregnant)
6. Breastfeeding
7. No nearby party for assistance if needed
8. Plans to go abroad or travel at more than 2 hours distance from Montreal during the trial period
9. Severe hypoglycemic episode within two weeks of screening or during the run-in period
10. Severe hyperglycemic episode requiring hospitalization in the last 3 months
11. Current use of glucocorticoid medication (except low stable dose and inhaled steroids)
12. Known or suspected allergy to the trial products
13. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator
14. Anticipation of a significant change in exercise regimen between admission and end of the trial (i.e. starting or stopping an organized sport)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Percentage of time of glucose levels spent between 3.9 and 10 mmol/L. | 288 hours

SECONDARY OUTCOMES:
Percentage of time of glucose levels spent between 3.9 and 7.8 mmol/L | 288 hours
Percentage of time of glucose levels spent below 3.9 mmol/L | 288 hours
Percentage of time of glucose levels spent below 3.3 mmol/L | 288 hours
Percentage of time of glucose levels spent below 2.8 mmol/L | 288 hours
Percentage of time of glucose levels spent above 10.0 mmol/L | 288 hours
Percentage of time of glucose levels spent above 13.9 mmol/L | 288 hours
Percentage of time of glucose levels spent above 16.7 mmol/L | 288 hours
Percentage of time of overnight glucose levels spent between 3.9 and 7.8 mmol/L | 72 hours
  The overnight period is between 00:00 and 06:00
Percentage of time of overnight glucose levels spent between 3.9 and 10.0 mmol/L | 72 hours
  The overnight period is between 00:00 and 06:00
Percentage of time of overnight glucose levels spent below 3.9 mmol/L | 72 hours
  The overnight period is between 00:00 and 06:00
Percentage of time of overnight glucose levels spent below 3.3 mmol/L | 72 hours
  The overnight period is between 00:00 and 06:00
Percentage of time of overnight glucose levels spent below 2.8 mmol/L | 72 hours
  The overnight period is between 00:00 and 06:00
Percentage of time of overnight glucose levels spent above 10.0 mmol/L | 72 hours
  The overnight period is between 00:00 and 06:00
Percentage of time of overnight glucose levels spent above 13.9 mmol/L | 72 hours
  The overnight period is between 00:00 and 06:00
Percentage of time of overnight glucose levels spent above 16.7 mmol/L | 72 hours
  The overnight period is between 00:00 and 06:00
Total number of hypoglycemic events below 3.1 mmol/L | 288 hours
Number of nights with hypoglycemic events below 3.1 mmol/L | 72 hours
Number of days with hypoglycemic events below 3.1 mmol/L | 126 hours
Mean glucose levels | 288 hours
Standard deviation of glucose levels | 288 hours
Time between failures due to glucose sensor unavailability | 288 hours
Coefficient of variation of glucose levels | 288 hours
Between-day variability in glucose levels | 288 hours
Total daily insulin dose | 24 hours
Standard deviation of insulin delivery | 288 hours
Coefficient of variation of insulin delivery | 288 hours
Between-day variability in insulin delivery | 288 hours
Total number of hours of glucose sensor availability | 288 hours
Percentage of time of glucose sensor availability | 288 hours
Time between failures due to pump connectivity | 288 hours
Percentage of time when patients switched back to insulin pump therapy | 288 hours
Number of hours when patients switched back to insulin pump therapy | 288 hours
Percentage of time when the closed-loop was automatically switched to insulin pump therapy | 288 hours
Number of hours when the closed-loop was automatically switched to insulin pump therapy | 288 hours
Number of days with at least one technical problem | 288 hours
Number of calls for technical issues related to the closed-loop system | 288 hours
Number of patients calling for technical issues related to the closed-loop system | 288 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (2):
- Canada (2):
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haidar A, Legault L, Raffray M, Gouchie-Provencher N, Jacobs PG, El-Fathi A, Rutkowski J, Messier V, Rabasa-Lhoret R. Comparison Between Closed-Loop Insulin Delivery System (the Artificial Pancreas) and Sensor-Augmented Pump Therapy: A Randomized-Controlled Crossover Trial. Diabetes Technol Ther. 2021 Mar;23(3):168-174. doi: 10.1089/dia.2020.0365. Epub 2020 Dec 31. PMID 33050728